CLINICAL TRIAL: NCT02558257
Title: Perception of the Palliative Care Encounter by Patients Who Are Referred to Outpatient Supportive/ Palliative Care
Brief Title: Perception of Palliative Care Encounter
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0578; NCI-2017-01598 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Survey; Questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative Care Survey: Initial consultation visit followed by phone survey within 1 week +/- 4 days of initial consultation.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Participants complete palliative care survey within 1 week +/- 4 days of initial consultation via phone survey conducted by Research nurse/assistant.
  Other Names: Questionnaire

SUMMARY:
Objectives:

Primary Objective The primary objective is to determine patients' perceptions of the timeliness of their referral to an outpatient palliative care clinic.

The secondary objectives are to determine:

1. The factors and variables associated with perception of timeliness such as age, gender, and symptom distress
2. The patients' perceptions of the physical environment of the outpatient clinic at UT MD Anderson Cancer Center (UTMDACC) such as lighting, music, and lack of a waiting room; and
3. If there is an association between level of distress (physical, psychological, and spiritual distress as measured by Edmonton Symptom Assessment Scale (ESAS) and the usefulness of the referral to palliative care center.

DETAILED DESCRIPTION:
If participant agrees to take part, they will complete 1 questionnaire over the phone, in person, or via e-mail about their first consultation experience, within 1 month after their visit. It should take about 15 minutes to complete. Health information about participant (such as their name, medical record number, telephone number, e-mail address, IP address, age, gender, race/ethnicity and cancer type) will also be collected but will not be shared with anyone outside of MD Anderson, except when required for regulatory purposes, or when required to be shared with study sponsors or study monitors. Participant's survey answers will not be shared with the Supportive Care staff.

Distress Plan:

Telephone - If participant experiences any distress while answering the survey questions, the research assistant will immediately contact our nurse in the Supportive Care Center. Participant will be contacted immediately to provide telephone counseling or address any other issue that may be causing distress. Our phone care nurse will offer participant to schedule a face-to-face visit with one of the Supportive Care physicians or to see a nurse in the Supportive Care Center.

In-person - If participant experiences significant and high levels of distress while participating in the study, we will refer participant to their primary care physician, physician in the Supportive Care Center or one of the supportive care counselors.

Online - If participant experiences significant and high levels of distress while completing the online survey, they may stop the survey and call the Supportive Care Center (during office hours) or the Supportive Care Mobile Team (after office hours or weekends). The contact information will be displayed on each page of the online survey.

Patient's participation on the study will be over after they have completed the questionnaire. Participant's de-identified study information will be kept by the Principal Investigator in a locked file cabinet and password protected electronic study database for 5 years after publication of the research and then destroyed. Online survey responses, demographics, e-mail address, and IP address will be stored indefinitely in a secured database by the Qualtrics team.

ELIGIBILITY:
Inclusion Criteria:

1. Have advanced cancer, defined as locally advanced, metastatic or incurable disease
2. >/=18 years of age
3. Seen at UTMDACC outpatient Supportive Care Center for consultation
4. Provided informed consent

Exclusion Criteria:

1. Memorial Delirium Assessment Scale (MDAS) >/= 13.
2. Inability to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have undergone a consultation with a supportive Care doctor in the Supportive Care Center at The University of Texas MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2015-08-16 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Participants' Perceptions of Timeliness of Referral to an Outpatient Palliative Care Clinic | 1 day
  Percentage of respondents who report that their referral to supportive care was late (including "late" and "too late") estimated with a standard error not larger than 0.04.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique N. Wong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org